CLINICAL TRIAL: NCT03139292
Title: Comparative Evaluation of Ambu AuraGain Laryngeal Mask and Proseal Laryngeal Mask Airway in Spontaneously Breathing Patients Undergoing Elective Surgery Under General Anaesthesia
Brief Title: Comparative Evaluation of Ambu AuraGain Laryngeal Mask and Proseal Laryngeal Mask Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Main Hospital (Other)
Responsible Party: Principal Investigator, Dr.Deb Sanjay Nag, Consultant, Tata Main Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201-26104-152-206580
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Laryngeal Masks

STUDY DESIGN:
Intervention Model Description: Prospective randomized single blinded parallel group controlled study
Who Masked: Participant, Outcomes Assessor
Masking Description: Sequentially numbered, sealed, opaque envelopes: Participant and Outcome Assessor Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ProSeal Laryngeal Mask Airway (Experimental): Intravenous (0.02mg/kg Midazolam and 2 microgram/kg Fentanyl) and oxygen via a face mask will be administered. Two minutes later, general anesthesia will be induced using 2 mg/kg intravenous Propofol mixed with 25 mg Lidocaine Injected over 30 seconds, Mask ventilation commence and continue for at least 30 seconds until conditions are suitable for PLMA insertion
  Interventions: Device: ProSeal Laryngeal Mask Airway
- AmbuAuraGain Laryngeal Mask Airway (Experimental): Intravenous (0.02mg/kg Midazolam and 2 microgram/kg Fentanyl) and oxygen via a face mask will be administered. Two minutes later, general anesthesia will be induced using 2 mg/kg intravenous Propofol mixed with 25 mg Lidocaine Injected over 30 seconds, Mask ventilation commence and continue for at least 30 seconds until conditions are suitable for AmbuAuraGain Laryngeal Mask Airway insertion
  Interventions: Device: AmbuAuraGain Laryngeal Mask Airway

INTERVENTIONS:
Device: ProSeal Laryngeal Mask Airway — ProSeal Laryngeal Mask Airway was used as the supraglottic device
  Arms: ProSeal Laryngeal Mask Airway
Device: AmbuAuraGain Laryngeal Mask Airway — AmbuAuraGain Laryngeal Mask Airway was used as the supraglottic device
  Arms: AmbuAuraGain Laryngeal Mask Airway

SUMMARY:
Comparison of two different supraglottic airway devices i.e., the ProSeal Laryngeal Mask Airway (PLMA) and Ambu AuraGain, a third generation laryngeal mask Airway.

DETAILED DESCRIPTION:
The study aims to compare the two devices with respect to:

Time taken for insertion. Insertion attempts or failed attempt. Oropharyngeal leak pressure Air leak Time taken to pass an orogastric tube Attempts to pass an orogastric tube or failed attempt. Haemodynamic variation Incidence of adverse events like failed insertion, aspiration-regurgitation, hypoxia (SpO2< 90%), bronchospasm, airway obstruction, gastric insufflation, coughing, gagging, retching, hiccup, coughing during removal, blood staining of the airway device and trauma to tongue, lip, teeth, or gums.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) Physical Status I & II
2. Patients undergoing limb or breast surgery
3. Patients undergoing elective surgery under general anesthesia and spontaneous ventilation.
4. Patients with expected duration of surgery of less than 2 hours.

Exclusion Criteria:

1. Patients with known or predicted difficult airway or Mallampati Grade (MPG) III or IV
2. Patients with mouth opening of less than 2.5 cm or cervical spine disease
3. Patients with H/o upper respiratory tract infection in the previous 10 days.
4. Patients with increased risk of regurgitation and aspiration (non-fasting patients, gastroesophageal reflux disease etc.)
5. Patients with a body mass index (BMI) > 30 kg/m2
6. Patients with past history of radiotherapy involving the hypopharynx/neck area 7Patients with expected duration of surgery of more than 2 hours.

8.Surgery to be performed to the head, neck or thorax, abdomen or in the lateral or prone positions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Success rate for the first attempt at insertion | 5 minutes
  A failed insertion attempt is defined as when removal of the device needed from the mouth.

SECONDARY OUTCOMES:
Time taken for insertion | 5 minutes
  Time taken for insertion from picking up the LMA till confirmation of effective ventilation
The number of insertion attempts | 5 minutes
  The number of insertion attempts or failed attempt to achieve effective ventilation. A failed insertion attempt is defined as when removal of the device needed from the mouth. Three attempts allowed before insertion will be considered a failure.
Intracuff and the oropharyngeal leak pressures after ensuring effective placement. | 5 minutes
  Intracuff and the oropharyngeal leak pressures after ensuring effective placement. These pressures will be determined by closing the expiratory valve of the circle system at a fresh gas flow of 3 l/min, note the airway pressure (maximum allowed: 40 cm H2O) at which equilibrium was reached.
The time taken for orogastric tube placement | 5 minutes
  The time taken for correct placement will be recorded, from Picking up the orogastric tube till confirmation of its placement.

CONTACTS AND LOCATIONS:
Locations (1):
- Tata Main Hospital, Jamshedpur, Jharkhand, India

IPD SHARING:
Plan to Share IPD: No